CLINICAL TRIAL: NCT06123793
Title: Assessment of Culprit-SYNTAX Score and No-reflow PIANO Score as Predictors of In-hospital and Short-term Clinical Outcomes in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Predictors of In-hospital and Short-term Clinical Outcomes in STEMI Patients Undergoing Primary PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ragab Kamel, Doctor, Assiut University
Other Study IDs: Predictors of outcomes in MI
Record Dates: First submitted 2023-09-20; First posted 2023-11-09 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess the culprit-SYNTAX score and no-reflow PIANO scores as possible predictors of in-hospital and short-term outcomes among patients with STEMI undergoing primary PCI

DETAILED DESCRIPTION:
ST-elevation myocardial infarction (STEMI) is the leading cause of death in cardiovascular patients. Percutaneous coronary intervention (PCI) is recommended as the preferred treatment for patients with STEMI. However, patients with (STEMI) undergoing primary (PCI) remain at high risk of adverse events, including death, reinfarction, stent thrombosis, and repeat revascularization. This underlines the need to identify predictors of impaired clinical outcomes in order to recognize higher-risk patients in the contemporary practice of primary PCI. STEMI patients show variable mortality risks, in order to assess individual risk, a number of mathematical models (scoring algorithms) have been developed as TIMI, GRACE 2.0, and ALPHA scores Similarly, angiographic scores were developed to assess the outcomes in STEMI patients, SYNTAX Score, has shown predictive value of in-hospital mortality among STEMI patients. Recently, the culprit-SYNTAX score appears to be as successful as the SYNTAX score in predicting stent thrombosis in patients with ACS and more successful in predicting 30-day deaths and major complications.

The no-flow phenomenon (NRP), one of the most common complications of primary PCI, significantly reduces the benefit of this procedure. The occurrence of NRP following PPCI leads to an unfavorable short-term prognosis by increasing the risk of complications and in some cases, of death. A new score system (the PIANO score) based on six clinical variables was constructed and validated, was variables to predict angiographic no-reflow in STEMI patients undergoing primary PCI, and very recently showed potential prognostic value in patients with AMI undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

Patients presented with 1st episode of STEMI and undergoing primary PCI. For 1 year duration.

-

Exclusion Criteria:

1. Patient with STEMI in which thrombolytic therapy was used.
2. Patient with a history of previous CABG surgery.
3. Patient with a history of previous PCI.
4. Patient with a history of previous STEMI.
5. Patients with myocardial infarction with non-obstructive coronary arteries (MINOCA)
6. Patient with spontaneous coronary artery dissection (SCAD).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include patients presenting to Assiut University Heart Hospital with STEMI and undergoing primary PCI, each patient will be followed up 3 months post-PCI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
no-reflow PIANO score as predictor of cumulative MACE | 3 months
  Assess the role of The PIANO ( PredIction of Angiographic NO-reflow ) score as a predictor of cumulative (in-hospital and short-term) MACE over 3 months period in STEMI patients undergoing primary PCI
  The PIANO score ranges from 0 - 14 and it predicts NO Reflow (a complication of PCI), patients with higher scores have a higher risk of developing NO Reflow as a complication
  The PIANO score depends on the following:
  * Age ≥70 years,( 2 points )
  * absence of pre-infarction angina ( 3 points )
  * total ischemic time ≥4 h ( 1 point )
  * left anterior descending as the culprit artery ( 1 point )
  * pre-PCI TIMI flow grade ≤1 ( 2 points ) pre-PCI TIMI thrombus score ≥4 ( 5 points )
  we will look if patients undergoing primary PCI with high PIANO scores will have a higher risk of poor outcomes.
culprit-SYNTAX score as predictor of cumulative MACE | 3 months
  SYNTAX score ( Synergy Between Percutaneous Coronary Intervention With Taxus and Cardiac Surgery) is a well-known score that assesses the severity and complexity of coronary artery disease and helps in choosing a treatment plan.
  - it ranges from 0 with no predefined maximum score, and it is calculated according to several angiographic parameters using this online calculator tool:https://syntaxscore.org/calculator/start.htm).
  the SYNTAX score can be calculated only for the culprit vessel ( culprit-SYNTAX) score
  we will look if patients undergoing primary PCI with high culprit-SYNTAX scores will have a higher risk of poor outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa R. Demitry, PhD, Study Director — Professor at cardiovascular medicine department , assiut university
Locations (1):
- Abdelrahman Ragab, Asyut, Egypt

REFERENCES:
- [Background] Tanik VO, Cinar T, Arugaslan E, Karabag Y, Hayiroglu MI, Cagdas M, Rencuzogullari I, Uluganyan M. The Predictive Value of PRECISE-DAPT Score for In-Hospital Mortality in Patients With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention. Angiology. 2019 May;70(5):440-447. doi: 10.1177/0003319718807057. Epub 2018 Oct 15. PMID 30322265
- [Background] Zijlstra F, Hoorntje JC, de Boer MJ, Reiffers S, Miedema K, Ottervanger JP, van 't Hof AW, Suryapranata H. Long-term benefit of primary angioplasty as compared with thrombolytic therapy for acute myocardial infarction. N Engl J Med. 1999 Nov 4;341(19):1413-9. doi: 10.1056/NEJM199911043411901. PMID 10547403
- [Background] Taniwaki M, Stefanini GG, Raber L, Brugaletta S, Cequier A, Heg D, Iniguez A, Kelbaek H, Serra A, Ostoijic M, Hernandez-Antolin R, Baumbach A, Blochlinger S, Juni P, Mainar V, Sabate M, Windecker S. Predictors of adverse events among patients undergoing primary percutaneous coronary intervention: insights from a pooled analysis of the COMFORTABLE AMI and EXAMINATION trials. EuroIntervention. 2015 Aug;11(4):391-8. doi: 10.4244/EIJY14M07_12. PMID 25042419
- [Background] Hizoh I, Domokos D, Banhegyi G, Becker D, Merkely B, Ruzsa Z. Mortality prediction algorithms for patients undergoing primary percutaneous coronary intervention. J Thorac Dis. 2020 Apr;12(4):1706-1720. doi: 10.21037/jtd.2019.12.83. PMID 32395313
- [Background] Ayca B, Akin F, Celik O, Cetin S, Sahin I, Gulsen K, Kalyoncuoglu M, Katkat F, Okuyan E, Dinckal MH. Does SYNTAX score predict in-hospital outcomes in patients with ST elevation myocardial infarction undergoing primary percutaneous coronary intervention? Kardiol Pol. 2014;72(9):806-13. doi: 10.5603/KP.a2014.0064. Epub 2014 Mar 27. PMID 24671913
- [Background] Peker T, Boyraz B. Short-Term Prognostic Value of the Culprit-SYNTAX Score in Patients with Acute Myocardial Infarction. J Cardiovasc Dev Dis. 2023 Jun 24;10(7):270. doi: 10.3390/jcdd10070270. PMID 37504526
- [Background] Ndrepepa G, Tiroch K, Fusaro M, Keta D, Seyfarth M, Byrne RA, Pache J, Alger P, Mehilli J, Schomig A, Kastrati A. 5-year prognostic value of no-reflow phenomenon after percutaneous coronary intervention in patients with acute myocardial infarction. J Am Coll Cardiol. 2010 May 25;55(21):2383-9. doi: 10.1016/j.jacc.2009.12.054. PMID 20488311
- [Background] Pantea-Rosan LR, Pantea VA, Bungau S, Tit DM, Behl T, Vesa CM, Bustea C, Moleriu RD, Rus M, Popescu MI, Turi V, Diaconu CC. No-Reflow after PPCI-A Predictor of Short-Term Outcomes in STEMI Patients. J Clin Med. 2020 Sep 12;9(9):2956. doi: 10.3390/jcm9092956. PMID 32932736
- [Background] Dai C, Liu M, Zhou Y, Lu D, Li C, Chang S, Chen Z, Qian J, Ge J. A score system to predict no-reflow in primary percutaneous coronary intervention: The PIANO Score. Eur J Clin Invest. 2022 Feb;52(2):e13686. doi: 10.1111/eci.13686. Epub 2021 Oct 11. PMID 34596236
- [Background] Dai C, Yang Z, Liu M, Zhou Y, Lu D, Chang S, Li C, Lu H, Chen Z, Qian J, Ge J. Prognostic value and clinical usefulness of PIANO score in patients undergoing primary percutaneous coronary intervention. Int J Cardiol. 2023 Nov 1;390:131258. doi: 10.1016/j.ijcard.2023.131258. Epub 2023 Aug 17. PMID 37574024